CLINICAL TRIAL: NCT04337255
Title: MIND Diet and Dementia Prevention in Ischemic Stroke Patients
Brief Title: Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet in Stroke Patients Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Chicago (Other); Advocate Hospital System (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Neelum T. Aggarwal, MD, Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18052104-IRB01
Record Dates: First submitted 2019-12-12; First posted 2020-04-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Decline; Dementia, Vascular; Alzheimer Disease; Dementia; Stroke
MeSH Terms: conditions — Cognitive Dysfunction; Dementia, Vascular; Alzheimer Disease; Dementia; Stroke

STUDY DESIGN:
Intervention Model Description: MIND diet intervention
Who Masked: Outcomes Assessor
Masking Description: Single ( Outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIND DIET intervention (Active Comparator): Allocation and blinding 3 year intervention of MIND Diet + counseling
  Interventions: Other: Behavioral Dietary intervention ( MIND Diet)
- Usual care diet intervention (Placebo Comparator): 3 year Intervention of usual care diet + counseling

INTERVENTIONS:
Other: Behavioral Dietary intervention ( MIND Diet) — The MIND diet is a hybrid of the Mediterranean and DASH diets but with selected modifications based on the most compelling evidence in the diet dementia field. The MIND diet has the same basic components of the DASH and Mediterranean diets, such as emphasis on natural plant based foods and limited animal and high saturated fat foods, but uniquely specifies green leafy vegetables and berries as well as food component servings that reflect the nutrition dementia evidence.
  Arms: MIND DIET intervention
Other: Behavioral Usual Care Diet Intervention — The Usual Care diet is comprised of both westernized (e.g. Steak, Mac n Cheese) and healthy ( veggie chili) food components

SUMMARY:
To test the effects of a 2- to 3-year intervention of the MIND diet versus usual post-stroke care on cognitive decline, the characteristic feature of dementia, and on brain biomarkers of Alzheimer's Disease (AD) and vascular disease in a Phase Ill randomized controlled trial of 250 patients hospitalized for acute ischemic stroke, aged 55 years or older, and without dementia who are discharged home following hospitalization.

DETAILED DESCRIPTION:
The Mediterranean-DASH diet intervention for Neurodegenerative Delay (MIND in Stroke patients is designed to test the effects of a 2-3 year intervention of a hybrid of the Mediterranean and DASH diets, called MIND on 250 older patients, without dementia who are hospitalized for acute stroke who are discharged home following hospitalization. The MIND diet has the same basic components of the DASH and Mediterranean diets, such as emphasis on natural plant based foods and limited animal and high saturated fat foods, but uniquely specifies green leafy vegetable and berries as well as food component servings that reflect the nutrition dementia evidence. In this study we will test the effects of a 2- to 3-year intervention of the MIND diet (3 months of delivered meals followed by dietary and general stroke health counseling) versus usual post-stroke care (3 months delivered self-selected meals followed by general stroke health counseling) on change on cognitive outcomes over 24 to 36 months. Biological effects of the MIND diet will be assessed by measurement of brain macro and microstructural integrity in all trial participants. Other biochemical markers will be assessed in the entire group of 250 participants including: plasma Abeta42/beta40, brain derived neurotropic factor (BDNF) and plasma markers of oxidative stress and inflammation. The trial will examine potential effect mediators and modifiers by a number of cardiovascular risk factors, AD biomarkers and biological mechanisms. The proposed study has 3 recruitment sites, Rush University Medical Center, University of Chicago, and Advocate Christ Hospital all located in Chicago.

ELIGIBILITY:
* Inclusion Criteria
* Men and women, 55 years of age - inclusive- or older
* Acute stroke as defined by an acute focal neurological deficit in combination with one of the following: acute ischemic infarct (stroke) as documented by either a DWl positive lesion on MR imaging or a new lesion on a delayed CT scan
* Written informed consent by patient prior to study participation
* Willingness to complete all assessments and participate in follow-up
* Willing to participate and give informed consent
* Adequate Visual and auditory acuity to undergo neuropsychological testing
* Exclusion criteria
* CDR>=0.5
* Nuts, berries, olive oil, or fish allergies
* Use of medications to treat Alzheimer's disease or Parkinson's disease
* Aphasia
* Conditions of psychosis or bipolar disorder judged by study investigators to potentially interfere with study compliance over 3 years
* Report of alcohol or substance abuse within six months, or heavy alcohol consumption (>2 drinks/d women; >3 drinks/d men)
* Unstable or recent onset of cardiovascular disease, such as myocardial infarction within six months or presence of congestive heart failure (Stages II-IV)
* Cancer treatment <= 5 years except non-melanoma skin cancer , basal cell skin cancer (this criterion may be waived at the site PI's discretion)
* Illness that might be associated with weight change, such as a history of stomach or gastrointestinal conditions (Inflammatory Bowel Disease, Crohn's Disease, malabsorption, colostomy, bowel resection, gastric bypass surgery, etc.)
* History of liver disease, HIV or Hepatitis C
* An intracerebral hemorrhage as documented on CT or MRI
* Pre- hospitalization diagnosis of dementia or mild cognitive impairment
* Patients presenting one of the following diseases: cerebral venous thrombosis, traumatic cerebral hemorrhage, intracerebral hemorrhage because of a known or image-guided assumed vascular malformation, pure meningeal or intraventricular hemorrhage
* Patients presenting a malignant disease with life expectancy < 3 years
* Residence in a nursing home and thus going back to nursing home upon discharge
* Participation in an ongoing investigational drug study
* Exception to these guidelines will be rare but may be considered on a case by case basis at the discretion of the PI's

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive score | 3-years
  3-year change in global cognitive score. The global cognitive score is a composite score, based on the average of z scores of the 19 individual tests scores, with a mean of 0 and standard deviation of 1. Higher scores reflect high global cognitive function.

SECONDARY OUTCOMES:
Change in brain MRI derived markers of macro and micro structural integrity (cubic Centimeters), total brain volume, hippocampal volume and white matter hyperintensity volume ( cubic centimeters) | 3-years
  130 participants total ( 65 in each treatment group)
Change in 5 individual cognitive domains | 3-years
  Change in 5 individual domains that include executive functioning, perceptual speed, episodic memory, semantic and working memory. Each domain is made up of atleast 2 cognitive tests that are z scored and averaged for that domain. Higher scores on each domain reflects higher cognition in that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Neelum T Aggarwal, MD., Principal Investigator — Rush University Medical Center; Christy Tangney, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Electronic data will be made available after trial completion
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months following publication of results
Access Criteria: Review & Approval by the Publications and Presentation Committee

REFERENCES:
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666
- [Background] Cherian L, Wang Y, Fakuda K, Leurgans S, Aggarwal N, Morris M. Mediterranean-Dash Intervention for Neurodegenerative Delay (MIND) Diet Slows Cognitive Decline After Stroke. J Prev Alzheimers Dis. 2019;6(4):267-273. doi: 10.14283/jpad.2019.28. PMID 31686099
- [Derived] Ventrelle J, Lukaszewicz B, Claysen M, Setia B, Aggarwal NT, Tangney CC; NOURISH Study Team. A framework for monitoring intervention fidelity: The NOURISH trial. Contemp Clin Trials. 2025 Nov;158:108104. doi: 10.1016/j.cct.2025.108104. Epub 2025 Oct 4. PMID 41052713